CLINICAL TRIAL: NCT01323790
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of NKTR-118 in Patients With Non-Cancer-Related Pain and Opioid-Induced Constipation (OIC)
Brief Title: Assessment of Efficacy and Safety in Patients With Non-cancer-related Pain and Opioid-induced Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3820C00005; 2011-001986-41 (EudraCT Number)
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Induced Constipation (OIC)
Keywords: Non-Cancer-Related Pain; Opioid-Induced Constipation
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naloxegol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Oral treatment
  Interventions: Drug: NKTR-118
- 2 (Experimental): Oral treatment
  Interventions: Drug: NKTR-118
- 3 (Placebo Comparator): Oral treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NKTR-118 — 12.5 mg oral tablet once daily
  Arms: 1
Drug: NKTR-118 — 25 mg oral tablet once daily
  Arms: 2
Drug: Placebo — Placebo to NKTR-118
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the effect and safety of NKTR-118 treatment of opioid-induced constipation in patients with non-cancer-related pain, including those patients that have inadequate response to laxative therapy (LIR).

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent prior to any study-specific procedures.
* Self-reported active symptoms of OIC at screening (<3 SBMs/week and experiencing ≥1 reported symptom of hard/lumpy stools, straining, or sensation of incomplete evacuation/anorectal obstruction in at least 25% of BMs over the previous 4 weeks); and Documented confirmed OIC (<3 SBMs/week on average over the 2-week OIC confirmation period.
* Receiving a stable maintenance opioid regimen consisting of a total daily dose of 30 mg to 1000 mg of oral morphine, or equianalgesic amount(s) of 1 or more other opioid therapies for a minimum of 4 weeks prior to screening for non-cancer-related pain with no anticipated change in opioid dose requirement over the proposed study period as a result of disease progression.
* Willingness to stop all laxatives and other bowel regimens including prune juice and herbal products throughout the 2-week OIC confirmation period and the 12-week treatment period, and to use only bisacodyl as rescue medication if a BM has not occurred within at least 72 hours of the last recorded BM.

Exclusion Criteria:

* Patients receiving Opioid regimen for treatment of pain related to cancer.
* History of cancer within 5 years from first study visit with the exception of basal cell cancer and squamous cell skin cancer.
* Medical conditions and treatments associated with diarrhea, intermittent loose stools, or constipation.
* Other issues to the gastrointestinal tract that could impose a risk to the patient.
* Pregnancy or lactation.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2011-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Sostek, Study Director — AstraZeneca
Locations (120):
- United States (68):
  - Research Site, Mobile, Alabama
  - Research Site, Pell City, Alabama
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Sun Lakes, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, North Little Rock, Arkansas
  - Research Site, Sherwood, Arkansas
  - Research Site, Chino, California
  - Research Site, La Jolla, California
  - Research Site, Lincoln, California
  - Research Site, Modesto, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Bradenton, Florida
  - Research Site, Delray Beach, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Springs, Florida
  - Research Site, Ocala, Florida
  - Research Site, Sanford, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Conyers, Georgia
  - Research Site, John's Creek, Georgia
  - Research Site, Peoria, Illinois
  - Research Site, Council Bluffs, Iowa
  - Research Site, Wichita, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Chestnut Hill, Massachusetts
  - Research Site, Watertown, Massachusetts
  - Research Site, Livonia, Michigan
  - Research Site, Saint Clair Shores, Michigan
  - Research Site, Florissant, Missouri
  - Research Site, Henderson, Nevada
  - Research Site, Freehold, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Willingboro, New Jersey
  - Research Site, Great Neck, New York
  - Research Site, Hartsdale, New York
  - Research Site, North Massapequa, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Morrisville, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bellevue, Ohio
  - Research Site, Downingtown, Pennsylvania
  - Research Site, Jenkintown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pottstown, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Milan, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Houston, Texas
  - Research Site, Hurst, Texas
  - Research Site, Marshall, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugarland, Texas
  - Research Site, Clinton, Utah
  - Research Site, St. George, Utah
  - Research Site, West Jordan, Utah
- Belgium (6):
  - Research Site, Edegem, Belgium
  - Research Site, Roeselare, Belgium
  - Research Site, Antwerp
  - Research Site, Leuven
  - Research Site, Moerkerke
  - Research Site, Mouscron
- Croatia (4):
  - Research Site, Bjelovar
  - Research Site, Osijek
  - Research Site, Susak
  - Research Site, Zagreb
- Czechia (4):
  - Research Site, Choceň
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Zlín
- Hungary (10):
  - Research Site, Baja
  - Research Site, Budapest
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Pusztaszer
  - Research Site, Sátoraljaújhely
  - Research Site, Szeged
  - Research Site, Szikszó
  - Research Site, Úrhida
  - Research Site, Zalaegerszeg
- Spain (12):
  - Research Site, Málaga, Andalusia
  - Research Site, Barcelona, Catalonia
  - Research Site, Centelles (barcelona), Catalonia
  - Research Site, L'Hospitalet de Llobregat, Catalu?a
  - Research Site, Vic, Catalu?a
  - Research Site, Fuenlabrada, Madrid
  - Research Site, Almería
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Santiago de Compostela
  - Research Site, Valencia
  - Research Site, Valladolid
- Sweden (4):
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Stockholm
  - Research Site, Vällingby
- United Kingdom (12):
  - Research Site, Ayrshire, AYR
  - Research Site, Chesterfield, Derby
  - Research Site, Derby, Derby
  - Research Site, Plymouth, Devon
  - Research Site, London, Gt Lon
  - Research Site, Royton, Lancashire
  - Research Site, Thornton-Cleveleys, Lancashire
  - Research Site, Norwich, Norflk
  - Research Site, Barry, S Glam
  - Research Site, Bath, Somer
  - Research Site, Glasgow, Strath
  - Research Site, Coventry, Warwks

REFERENCES:
- [Derived] Lawson R, King F, Marsh K, Altincatal A, Cimen A. Impact of Treatment with Naloxegol for Opioid-Induced Constipation on Patients' Health State Utility. Adv Ther. 2016 Aug;33(8):1331-46. doi: 10.1007/s12325-016-0365-y. Epub 2016 Jun 24. PMID 27342744
- [Derived] Tack J, Lappalainen J, Diva U, Tummala R, Sostek M. Efficacy and safety of naloxegol in patients with opioid-induced constipation and laxative-inadequate response. United European Gastroenterol J. 2015 Oct;3(5):471-80. doi: 10.1177/2050640615604543. PMID 26535126
- [Derived] Chey WD, Webster L, Sostek M, Lappalainen J, Barker PN, Tack J. Naloxegol for opioid-induced constipation in patients with noncancer pain. N Engl J Med. 2014 Jun 19;370(25):2387-96. doi: 10.1056/NEJMoa1310246. Epub 2014 Jun 4. PMID 24896818
- See also: Clinical Study Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1852&filename=Clinical_Study_Protocol_redacted_D3820C00005.pdf
- See also: Clinical_Study_Report_Synopsis_D3820C00005 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1852&filename=Clinical_Study_Report_Synopsis_D3820C00005.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted in Belgium, Croatia, Czech Republic, Hungary, Spain, Sweden, United Kingdom, and the United States between 28 March 2011 and 20 September 2012.
Pre-assignment Details: The study duration was up to 18 weeks, consisting of an initial screening period lasting up to 2 weeks, a 2-week OIC confirmation period, during which the diagnosis of OIC and stability of the opioid regimen were confirmed, a 12-week treatment period, and a follow-up visit 2 weeks after the last dose of study drug.
Groups:
- NKTR-118 12.5 mg: NKTR-118 12.5 QD, oral treatment
- NKTR-118 25 mg: NKTR-118 25 mg QD, oral treatment
- Placebo: Placebo QD, oral treatment
Period: Overall Study
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Started | 233 | 234 | 233
Completed | 178 | 174 | 188
Not Completed | 55 | 60 | 45
Not completed — Other | 3 | 2 | 1
Not completed — Lost to Follow-up | 11 | 9 | 9
Not completed — Study-Specific Withdrawal Criteria | 0 | 3 | 3
Not completed — Lack of Efficacy | 3 | 0 | 3
Not completed — Adverse Event | 11 | 24 | 12
Not completed — Eligibility Criteria Not Fulfilled | 0 | 0 | 1
Not completed — Withdrawal by Subject | 23 | 20 | 13
Not completed — Did Not Receive Treatment | 2 | 0 | 1
Not completed — Severe non-compliance with protocol | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Population: A total of 4 patients (2 patients in the NKTR-118 25 mg and 1 patient each in the NKTR-118 12.5 mg and placebo groups) had been previously randomized within the NKTR-118 program at a different study center. These patients were excluded from the ITT and Safety analysis sets. Baseline characteristics are summarized based on the ITT analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo | Total
Number analyzed (Participants) | 232 | 232 | 232 | 696
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.0 (11.02) | 51.9 (12.11) | 52.3 (11.62) | 52.1 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 147 | 145 | 441
  Male | 83 | 85 | 87 | 255
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2 | 4
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 41 | 40 | 44 | 125
  White | 187 | 189 | 183 | 559
  Other | 2 | 1 | 3 | 6
Baseline laxative response status [Number; unit: Participants] — Laxative response status was determined at the screening visit (Visit 1) based on the Baseline Laxative Response Status Questionnaire. Patients were classified as: Laxative Inadequate Responder (LIR: patients who reported moderate, severe, or very severe symptoms in at least 1 of the 4 stool symptom domains); Laxative Adequate Responder (LAR: patients who reported no symptoms or only mild symptoms); and Laxative Unknown Responder (LUR: patients who had not taken laxatives over the previous 2 weeks or who had taken 1 or more laxative classes on <4 days over the previous 2 weeks).
  Participants
    Laxative Inadequate Response (LIR) | 125 | 124 | 121 | 370
    Laxative Adequate Response (LAR) | 5 | 5 | 4 | 14
    Laxative Unknown Response (LUR) | 102 | 103 | 107 | 312

OUTCOME MEASURES:

1. Primary Outcome: Response (Responder/Non-responder) to Study Drug During Weeks 1 to 12
Description: Responder was defined as having at least 3 spontaneous bowel movements (SBMs)/week with at least 1 SBM/week increase over baseline for at least 9 out of the 12 treatment weeks and 3 out of the last 4 treatment weeks during the double-blind treatment period. An SBM is a bowel movement occurring 24 hours or more since the last use of rescue medication.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: The ITT analysis set included all randomized patients, with the exception of patients who were found to have randomized multiple times within the program at different centers.
Measure: Number; unit: Number of patients
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 232 | 232 | 232
Number of patients | 81 | 92 | 68
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; Analysis via Cochran Mantel-Haenszel test stratified by response to laxatives at baseline (LIR, LAR, LUR); Test type: Superiority or Other; p = 0.202, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.188, 95% CI 2-sided [0.911 to 1.548]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; Analysis via Cochran Mantel-Haenszel test stratified by response to laxatives at baseline (LIR, LAR, LUR); Test type: Superiority or Other; p = 0.021, Cochran-Mantel-Haenszel; Risk Ratio (RR) = 1.348, 95% CI 2-sided [1.045 to 1.739]

2. Secondary Outcome: Response (Responder/Non-responder) to Study Drug in the LIR Subgroup During Weeks 1 to 12
Description: Responder is defined as having at least 3 SBMs/week, with at least 1 SBM/week increase over baseline for at least 9 out of 12 weeks and at least 3 out of the last 4 weeks.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: The ITT analysis set included all randomized patients, with the exception of patients who were found to have randomized multiple times within the program at different centers. The LIR subgroup used 1 or more laxative classes for at least 4 days in the 2 weeks prior to entry and reported moderate to very severe symptoms.
Measure: Number; unit: Number of patients
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 125 | 124 | 121
Number of patients | 53 | 58 | 38
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; Test type: Superiority or Other; p = 0.074, Cochran-Mantel-Haenszel — Response rate over Weeks 1 to 12 in the LIR subgroup is a key secondary endpoint included in the multiple testing procedure; Risk Ratio (RR) = 1.350, 95% CI 2-sided [0.967 to 1.884]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; Test type: Superiority or Other; p = 0.014, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Risk Ratio (RR) = 1.489, 95% CI 2-sided [1.078 to 2.058]

3. Secondary Outcome: Time (in Hours) to First Post-dose Laxation Without the Use of Rescue Laxatives Within the Previous 24 Hours
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 232 | 232 | 232
Hours | 19.3 [9.4 to 22.3] | 12.0 [7.0 to 21.5] | 37.2 [30.0 to 46.9]

4. Secondary Outcome: Change From Baseline in Mean Number of Days Per Week With at Least 1 SBM During Weeks 1 to 12
Time Frame: 12 weeks
Population: The ITT analysis set included all randomized patients who had evaluable data at baseline and post-baseline, with the exception of patients who were found to have randomized multiple times within the program at different centers.
Measure: Least Squares Mean (Standard Error); unit: Number of Days
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 228 | 226 | 231
Number of Days | 2.12 (0.12) | 2.41 (0.13) | 1.73 (0.12)
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; Analysis via Mixed Model Repeated Measures (MMRM) with fixed effects for baseline, baseline laxative response, treatment and treatment time interaction. Study pooled center is included as a random effect; Test type: Superiority or Other; p = 0.010, Mixed Models Analysis; LS mean difference = 0.39, 95% CI 2-sided [0.09 to 0.69]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; Analysis via MMRM with fixed effects for baseline, baseline laxative response, treatment and treatment time interaction. Study pooled center is included as a random effect; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Ls mean difference = 0.68, 95% CI 2-sided [0.37 to 0.98]

5. Secondary Outcome: Change From Baseline in Degree of Straining
Description: A single-item straining question was asked via the eDiary: "How much did you strain during your bowel movement?" Patients responded on a 5 point Likert scale: 1=Not at all; 2=A little bit; 3=A moderate amount; 4=A great deal; 5=An extreme amount. A negative change from baseline indicates improvement.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 228 | 226 | 231
units on a scale | -0.67 (0.06) | -0.80 (0.06) | -0.48 (0.06)
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; Analysis via MMRM with fixed effects for baseline, baseline laxative response (LIR, non-LIR), treatment and treatment time interaction. Study pooled center is included as a random effect; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; LS mean difference = -0.19, 95% CI 2-sided [-0.32 to -0.06]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS mean difference = -0.32, 95% CI 2-sided [-0.45 to -0.18]

6. Secondary Outcome: Change From Baseline in Stool Consistency (Bristol Stool Scale)
Description: Patients rated stool consistency through completion of the BSS after each BM. The 7 stool types are: 1. Separate hard lumps, like nuts (hard to pass); 2. Sausage-shaped, but lumpy; 3. Like sausage, but with cracks on its surface; 4. Like a sausage or snake, smooth and soft; 5. Soft blobs with clear cut edges (passed easily); 6. Fluffy pieces with ragged edges, a mushy stool; 7. Watery, no solid pieces. A positive change from baseline indicates improvement.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 228 | 226 | 231
units on a scale | 0.54 (0.07) | 0.71 (0.07) | 0.26 (0.06)
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; LS mean difference = 0.28, 95% CI 2-sided [0.12 to 0.45]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS mean difference = 0.45, 95% CI 2-sided [0.29 to 0.62]

7. Secondary Outcome: Change From Baseline in Percent Numbers of Days With a CSBM (Complete Spontaneous Bowel Movement)
Description: A single-item question on the completeness of evacuation, developed and validated through 1:1 interviews with OIC patients, was asked via the eDiary: "Did you feel like your bowels were completely empty after the bowel movement?" Patients provided a yes or a no response. A positive change from baseline indicates improvement.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Percent days/week
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 228 | 226 | 231
Percent days/week | 23.48 (1.88) | 27.20 (1.93) | 16.76 (1.86)
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; LS mean difference = 6.72, 95% CI 2-sided [2.37 to 11.06]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS mean difference = 10.43, 95% CI 2-sided [6.03 to 14.84]

8. Secondary Outcome: Change From Baseline in Mean Spontaneous Bowel Movements/Week
Description: The number of spontaneous bowel movements/week was determined from the patient's eDiary.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Number of SBMs/week
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 228 | 226 | 231
Number of SBMs/week | 2.62 (0.18) | 3.14 (0.19) | 2.10 (0.18)
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.028, Mixed Models Analysis; LS mean difference = 0.52, 95% CI 2-sided [0.06 to 0.98]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS mean difference = 1.04, 95% CI 2-sided [0.58 to 1.51]

9. Secondary Outcome: Time (in Hours) to First Post-dose Laxation Without the Use of Rescue Laxatives Within the Previous 24 Hours in the Laxative Inadequate Response (LIR) Subgroup
Description: Time to first post-dose laxation without the use of rescue laxatives within the last 24 hours was calculated in hours as: Date/Time of first post-dose laxation without rescue - First dose date/time.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 125 | 124 | 121
hours | 12.8 [6.4 to 21.9] | 18.1 [6.5 to 22.8] | 38.2 [28.9 to 57.4]

10. Secondary Outcome: Change From Baseline in Patient Assessment of Constipation Symptoms Questionnaire (PAC-SYM)
Description: The PAC-SYM questionnaire is a 12-item questionnaire that evaluates the severity of symptoms of constipation in 3 domains (stool, rectal, and abdominal symptoms) on a 5-point Likert scale ranging from 0 (absent) to 4 (very severe) in the 2 weeks (14 days) prior to assessment. Each domain score is the mean of the non-missing items for that domain. The total score is the mean of all non-missing items (ie, symptoms). The range of the domain or total score is 0 (response is 'absent' for each item) to 4 (response is 'very severe' for each item). A negative change from baseline indicates improvement.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: The ITT analysis set included all randomized patients who had evaluable data at baseline and post-baseline, with the exception of patients who randomized multiple times at different centers. MMRM analysis includes all patients with baseline and at least 1 post-baseline assessment, while the Ns at Week 12 reflect patients providing data at Week 12.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 173 | 165 | 184
units on a scale
  Total score | -0.75 (0.05) | -0.81 (0.05) | -0.63 (0.05)
  Abdominal symptoms subscore | -0.67 (0.06) | -0.62 (0.06) | -0.72 (0.06)
  Rectal symptoms subscore | -0.59 (0.05) | -0.71 (0.05) | -0.47 (0.05)
  Stool symptoms subscore | -0.93 (0.07) | -1.04 (0.07) | -0.66 (0.07)
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.080, Mixed Models Analysis — Analysis for change in PAC-SYM total score from baseline (Week 1) to end of treatment (Week 12); LS mean difference = -0.12, 95% CI 2-sided [-0.26 to 0.01]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis — Analysis for change in PAC-SYM total score from baseline (Week 1) to end of treatment (Week 12); LS mean difference = -0.18, 95% CI 2-sided [-0.32 to -0.04]
Statistical Analysis 3: Comparison: NKTR-118 12.5 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.552, Mixed Models Analysis — Analysis for change in PAC-SYM abdominal symptoms subscore from baseline (Week 1) to end of treatment (Week 12); Slope = 0.05, 95% CI 2-sided [-0.11 to 0.20]
Statistical Analysis 4: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.236, Mixed Models Analysis — Analysis for change in PAC-SYM abdominal symptoms subscore from baseline (Week 1) to end of treatment (Week 12); LS mean difference = 0.09, 95% CI 2-sided [-0.06 to 0.25]
Statistical Analysis 5: Comparison: NKTR-118 12.5 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.095, Mixed Models Analysis — Analysis for change in PAC-SYM rectal symptoms subscore from baseline (Week 1) to end of treatment (Week 12); LS mean difference = -0.11, 95% CI 2-sided [-0.24 to 0.02]
Statistical Analysis 6: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Analysis for change in PAC-SYM rectal symptoms subscore from baseline (Week 1) to end of treatment (Week 12); LS mean difference = -0.24, 95% CI 2-sided [-0.37 to -0.10]
Statistical Analysis 7: Comparison: NKTR-118 12.5 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis — Analysis for change in PAC-SYM stool symptoms subscore from baseline (Week 1) to end of treatment (Week 12); LS mean difference = -0.27, 95% CI 2-sided [-0.44 to -0.10]
Statistical Analysis 8: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Analysis for change in PAC-SYM stool symptoms subscore from baseline (Week 1) to end of treatment (Week 12); LS mean difference = -0.38, 95% CI 2-sided [-0.56 to -0.21]

11. Secondary Outcome: Change From Baseline in Patient Assessment of Constipation Quality of Life (PAC-QOL) Satisfaction Domain
Description: The PAC-QOL scale is a 28-item self-report instrument designed to evaluate the burden of constipation on patients' everyday functioning and well-being in the 2 weeks (14 days) prior to assessment. Each item is rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely). The instrument can be used to generate an overall score, but is also reported to assess 4 specific constipation-related domains including: 1) Worries and concerns (11 items), 2) Physical discomfort (4 items), 3) Psychosocial discomfort (8 items), and 4) Satisfaction (5 items). Each domain score is the mean of the non-missing items for that domain. The total score is the mean of all non-missing items. The range of the domain or total score is 0 (response is 'not at all' for each item) to 4 (response is 'extremely' for each item). A negative change from baseline indicates improvement.
Time Frame: Baseline (Week 1) to end of treatment (Week 12)
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Number analyzed (Participants) | 168 | 167 | 185
units on a scale | -1.12 (0.09) | -1.30 (0.09) | -0.81 (0.09)
Statistical Analysis 1: Comparison: NKTR-118 12.5 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.011, Mixed Models Analysis; LS mean difference = -0.31, 95% CI 2-sided [-0.54 to -0.07]
Statistical Analysis 2: Comparison: NKTR-118 25 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS mean difference = -0.49, 95% CI 2-sided [-0.73 to -0.25]

ADVERSE EVENTS:
Description: Adverse Events are reported for those subjects who were randomized and receieved at least one dose of study treatment.
Arm/Group | NKTR-118 12.5 mg | NKTR-118 25 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 14/230 | 8/232 | 12/231
Other Adverse Events (participants affected / at risk) | 90/230 | 112/232 | 73/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-118 12.5 mg (N=230) | NKTR-118 25 mg (N=232) | Placebo (N=231)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
POST LAMINECTOMY SYNDROME (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
CHEST X-RAY ABNORMAL (Investigations) | 0 (0) | 0 (0) | 1 (1)
CSF CULTURE POSITIVE (Investigations) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
APHASIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
GRAND MAL CONVULSION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ALCOHOL ABUSE (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
ACCELERATED HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
MALIGNANT HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKTR-118 12.5 mg (N=230) | NKTR-118 25 mg (N=232) | Placebo (N=231)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4 (4) | 6 (6) | 5 (5)
ABDOMINAL PAIN (Gastrointestinal disorders) | 27 (27) | 44 (44) | 18 (18)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 (5) | 6 (6) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 19 (19) | 21 (21) | 10 (10)
FLATULENCE (Gastrointestinal disorders) | 4 (4) | 14 (14) | 7 (7)
NAUSEA (Gastrointestinal disorders) | 16 (16) | 20 (20) | 11 (11)
VOMITING (Gastrointestinal disorders) | 8 (8) | 16 (16) | 9 (9)
FATIGUE (General disorders) | 3 (3) | 6 (6) | 3 (3)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 7 (7) | 1 (1)
SINUSITIS (Infections and infestations) | 3 (3) | 7 (7) | 4 (4)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (4) | 6 (6) | 6 (6)
FALL (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 3 (3)
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 6 (6) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 12 (12) | 12 (12) | 4 (4)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7) | 1 (1)
DIZZINESS (Nervous system disorders) | 8 (8) | 3 (3) | 6 (6)
HEADACHE (Nervous system disorders) | 12 (12) | 12 (12) | 8 (8)
ANXIETY (Psychiatric disorders) | 5 (5) | 3 (3) | 4 (4)
HYPERTENSION (Vascular disorders) | 1 (1) | 8 (8) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days